CLINICAL TRIAL: NCT06452966
Title: The Impact and Effect of Traditional Chinese Medicine Treatment on Organ Failure in Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC3-052
Record Dates: First submitted 2024-05-20; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Organ Failure, Multiple; Indigestion; Delayed Gastric Emptying; Respiratory Failure; Morality
Keywords: acupuncture; chinese medicine; Organ Failure; intensive care
MeSH Terms: conditions — Multiple Organ Failure; Dyspepsia; Gastroparesis; Respiratory Insufficiency | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: a non-randomized real world data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Experimental): patients in the group will recived one of or a combination of the following intervantions:
  1. Oral Chinese medicine decoction:
     The Chinese medicine practitioner will personally examine the patient and judge the patient's condition through the four diagnostic methods of traditional Chinese medicine(TCM): sight, smell, inquiry, and incision. Based on the syndrome differentiation and treatment of the patient's condition, he or she will prescribe an oral Chinese herbal decoction, two to three times a day, for two weeks.
  2. Acupuncture or low level laser acupuncture treatment:
  Chinese medicine practitioners select acupuncture points for treatment based on the patient's condition and treat them twice a week for 20 minutes each time for a total of two weeks.
  the intervantion depents on the TCM doctor decision based on the patient's diagnosis and needs.
  in addition, the patients will recive ICU care and medication based on patient's needs.
  Interventions: Other: traditional Chinese medicine
- control group (Active Comparator): the patients in this group will receive routine ICU care. the patients will be recruted during the study period. the patients will not recive TCM intervantions.
  Interventions: Other: Routine ICU care
- Historical control (Other): Patients admitted to the same ICU in the period of 01.2019 to 12.2023. the patients did not recivied TCM intervantions
  Interventions: Other: historical Routine ICU care

INTERVENTIONS:
Other: traditional Chinese medicine — patients in the group will receive one of or a combination of the following interventions:
  Oral Chinese medicine decoction:
  The Chinese medicine practitioner will personally examine the patient and judge the patient's condition through the four diagnostic methods of traditional Chinese medicine(TCM): sight, smell, inquiry, and incision. Based on the syndrome differentiation and treatment of the patient's condition, he or she will prescribe an oral Chinese herbal decoction, two to three times a day, for two weeks.
  Acupuncture or low level laser acupuncture treatment:
  Chinese medicine practitioners select acupuncture points for treatment based on the patient's condition and treat them twice a week for 20 minutes each time for a total of two weeks.
  the intervantion depents on the TCM doctor decision based on the patient's diagnosis and needs.
  in addition, the patients will recive ICU care and medication based on patient's needs.
  Other Names: Oral Chinese medicine decoction and/or Acupuncture or low level laser acupuncture
  Arms: intervention group
Other: Routine ICU care — Patients will receive ICU care
  Other Names: ICU care
  Arms: control group
Other: historical Routine ICU care — Patients had received ICU care
  Other Names: Routine ICU care
  Arms: Historical control

SUMMARY:
Critically ill patients are at risk of or suffering from one or more key organs or organ system failure. This study will measure the effect of traditional Chinese medicine(TCM) interventions on critically ill patients admitted to the intensive care unit (ICU).

The goal of this clinical trial is to learn if traditional Chinese medicine(TCM) is effective for prevention and treatment of organ failure in ICU patients. Patients in this group will receive intervention for 2 weeks.

A multi-center non-randomized real word data study, will include 3 groups: intervention group (TCM)(n=70), control group and historical control group (admitted to the same ICU in the period of 01.2019 to 12.2023).

Main outcomes include sequential organ failure assessment (SOFA) score, ICU length of stay, hospital length of stay, number of days of respirator uses and western medicine medication used study follow up will be 2 weeks.

DETAILED DESCRIPTION:
Critically ill patients are at risk of or suffering from one or more key organs or organ system failure. This study will measure the effect of traditional Chinese medicine(TCM) interventions on critically ill patients admitted to the intensive care unit (ICU).

A multi center non-randomized real word data study, will include 3 groups: intervention group (n=70), control group (patients recruited enrolled to the ICU during the study period) and historical control group (admitted to the same ICU in the period of 01.2019 to 12.2023). The intervention group will receive traditional Chinese herbal medicine and/or acupuncture and/or low level laser applied on acupuncture points depending on TCM doctor decision and patient TCM diagnosis. Intervention period will be 2 weeks.

Main outcomes include sequential organ failure assessment (SOFA) score, ICU length of stay, hospital length of stay, number of days of respirator uses and western medicine medication used study follow up will be 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and above
* Surgical ICU patients
* The use of Chinese medicine must be approved by the attending physician in the surgical intensive care unit

Exclusion criteria:

* Patients' family members refuse TCM intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Intensive care unit length of stay | "through study completion, an average of 3 months".
  the number of days a patient stays in the Intensive care unit
hospital length of stay | "through study completion, an average of 3 months".
  The number of days a patient stays in the hospital
Mechanical ventilation time | "through study completion, an average of 3 months".
  The number of days a patient requires mechanical ventilation
Respiratory care center stay | "through study completion, an average of 3 months".
  The number of days a patient stays in the respiratory care center
Patient survival and mortality | "through study completion, an average of 1 year".
  Measure ICU, RCC, and hospital mortality

SECONDARY OUTCOMES:
Kidney function | baseline, day 1-14 of the study
  Measured by blood urea nitrogen (BUN)
Creatinine (creatinine) | baseline, day 1-14 of the study
  Creatinine (creatinine) levels in blood sample
Daily urine output | baseline, day 1-14 of the study
  Daily urine output in ml
Number of days out of the first 14 days the patients reach 70% of their target energy expenditure. | baseline, day 1-14 of the study
  Daily intake Number of days out of the first 14 days the patients reach 70% of their target energy expenditure.
Number of days to reach 80% of target energy expenditure. | baseline, day 1-14 of the study
  Daily intake, number of days out of the first 14 days the patients reach 80% of target energy expenditure.
Number of days to reach 100% of target energy expenditure. | baseline, day 1-14 of the study
  Daily intake Number of days out of the first 14 days the patients reach100% of target energy expenditure.
Oxygenation index | baseline, day 1-14 of the study
  FiO2 rate in ventilator
PaO2 rate | baseline, day 1-14 of the study
  patients PaO2 rate in ventilator
Respirator parameters | baseline, day 1-14 of the study
  Tidal volume (VT) in ventilator
Positive end-expiratory pressure (PEEP) | baseline, day 1-14 of the study
  Positive end-expiratory pressure (PEEP) in ventilator
Respiratory rate (RR) | baseline, day 1-14 of the study
  Respiratory rate (RR) in ventilator
Inspiratory airflow (V') | baseline, day 1-14 of the study
  Inspiratory airflow (V') in ventilator
Alanine transaminase (ALT) | baseline, day 1-14 of the study
  Alanine transaminase (ALT) levels in blood sample
Liver function | baseline, day 1-14 of the study
  Aspartate transaminase (AST) levels in blood sample
Alkaline phosphatase (ALP), | baseline, day 1-14 of the study
  Alkaline phosphatase (ALP), levels in blood sample
Albumin | baseline, day 1-14 of the study
  Albumin levels in blood sample
total protein | baseline, day 1-14 of the study
  total protein levels in blood sample
Bilirubin, | baseline, day 1-14 of the study
  Bilirubin, levels in blood sample
L-lactate dehydrogenase (LD) | baseline, day 1-14 of the study
  L-lactate dehydrogenase (LD) levels in blood sample
Prothrombin time (PT) | baseline, day 1-14 of the study
  Prothrombin time (PT)
Cardiovascular function | baseline, day 1-14 of the study
  Measured by blood pressure
use of vasopressors. | baseline, day 1-14 of the study
  Measured by use of vasopressors.
Glasgow Coma Scale (GCS) | baseline, day 1-14 of the study
  Glasgow Coma Scale (GCS)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan